CLINICAL TRIAL: NCT04973943
Title: Donor-derived Cell Free DNA as a Potential New Biomarker in Cardiac Transplantation: Role in Acute Rejection
Brief Title: Donor-derived Cell Free DNA as a New Biomarker in Cardiac Acute Rejection
Acronym: FreeDNA-CAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Javier Segovia Cubero, Head of Cardiology Department, Puerta de Hierro University Hospital
Other Study IDs: FreeDNA-CAR
Record Dates: First submitted 2021-03-15; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Heart Transplant Rejection
Keywords: Donor-derived cell Free DNA; Acute cellular rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Donor-derived cell Free DNA — Measurement of dd-cfDNA and comparison against grade of rejection as determined by endomyocardial biopsy, taken simultaneously

SUMMARY:
FreeDNA-CAR is a prospective, observational multicenter study, that will include a total of 200 adult heart transplant (HT) patients from 14 centers in Spain. Our main objective is to test donor-derived Cell-Free DNA (dd-cfDNA) against endomyocardial biopsy (EMB) for the diagnosis of acute cellular rejection.

DETAILED DESCRIPTION:
All patients will be enrolled immediately after HT, and will undergo undergo routine surveillance EMB at 15 days, 1 month, 2, 3, 4, 6 and 12 months after HT. Simultaneously with each EMB, dd-cfDNA will be measured in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old who undergo heart transplant during the recruiting period

Exclusion Criteria:

* Patients with moderate or severe Primary Graft Dysfunction
* Patients on invasive mechanical ventilation 15 days after heart transplant
* Patients on renal replacement therapy, continuous or periodic, 15 days after heart transplant
* Heart Transplant due to a cardiomyopathy that could potentially recur on the graft (cardiac amyloidosis, Chagas disease or sarcoidosis, amongst others)
* Multiorgan transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant recipients aged 18 and over
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Association between dd-cfDNA levels and the presence of acute cellular rejection | 1 year
  Association between dd-cfDNA levels above a certain cut-point and the presence of treatable acute cellular rejection as determined by endomyocardial biopsy (graded by International Society of Heart and Lung Transplantation 2010 classification, grade > 1R).

SECONDARY OUTCOMES:
Area under curve for dd-cfDNA | 1 year
  To define a cutt-off point of dd-cfDNA level with a high negative predictive value that could obviate the need to perform surveillance endomyocardial biopsies
Correlation between dd-cfDNA and antibody mediated rejection (AMR) | 1 year
  Correlation between dd-cfDNA and antibody mediated rejection (AMR)
Association between dd-cfDNA and immunosuppressive (IS) treatment | 1 year
  Subanalysis of association between dd-cfDNA and rejection stratified by IS regimen (type and dose of drug).
Association between dd-cfDNA (%) and left ventricular ejection fraction | 1 year
  Association between dd-cfDNA and left ventricular ejection fraction (LVEF). All echocardiograms will be performed on the same day of EMB.
Determine the biomarker's kinetics at 15 days post-transplant | 15 days
  Determine dd-cfDNA levels at 15 days post-transplant in absence of rejection
Association between dd-cfDNA levels and cytomegalovirus (CMV) infection | 1 year
  Association between dd-cfDNA levels and CMV infection as determined by CMV polymerase chain reaction (number of copies per ml)
Determine a cut-off point of dd-cfDNA that allows to differentiate between acute cellular rejection (ACR) and antibody mediated rejection (AMR) | 1 year
  Determine a cut-off point of dd-cfDNA that allows to differentiate between acute cellular rejection (ACR) and antibody mediated rejection (AMR)

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - University Hospital Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Bellvitge, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital 12 octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Virgen del Rocio, Seville
  - Hospital La Fe, Valencia

REFERENCES:
- [Derived] Jimenez-Blanco M, Crespo-Leiro MG, Garcia-Cosio Carmena MD, Gomez Bueno M, Lopez-Vilella R, Ortiz-Bautista C, Farrero-Torres M, Zegri-Reiriz I, Diaz-Molina B, Garcia-Romero E, Rangel-Sousa D, Salterain N, Garrido Bravo I, Segovia-Cubero J. Donor-derived cell-free DNA as a new biomarker for cardiac allograft rejection: A prospective study (FreeDNA-CAR). J Heart Lung Transplant. 2025 Apr;44(4):560-569. doi: 10.1016/j.healun.2024.11.009. Epub 2024 Nov 20. PMID 39577511